CLINICAL TRIAL: NCT02366884
Title: Atavistic Chemotherapy and Immunotherapy in Advanced, Metastatic, and Otherwise Incurable and Lethal Cancers Under Conventional Treatments
Brief Title: Clinical Evaluation of a New Form of Cancer Therapy (Atavistic Chemotherapy) Based on the Principles of Atavistic Metamorphosis (2011)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Frank Arguello Cancer Clinic (Industry)
Collaborators: Instituto de Ciencia y Medicina Genomica, Torreon, Coah. Mexico www.institutodeciencia.com (Unknown)
Responsible Party: Principal Investigator, Frank Arguello, MD, Director, Dr. Frank Arguello Cancer Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACI/2015
Record Dates: First submitted 2015-02-09; First posted 2015-02-19 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Neoplasms
Keywords: malignant; atavistic chemotherapy; cancer
MeSH Terms: conditions — Neoplasms | interventions — Anti-Bacterial Agents; Antifungal Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anti-bacterial agents (Experimental): Combination of two selected anti-bacterial agents with documented anti-cancer properties
  Interventions: Drug: Anti-Bacterial Agents
- Anti-fungal agents (Experimental): Combination of two selected anti-fungal agents with documented anti-cancer properties
  Interventions: Drug: Anti-Fungal Agents
- Anti-protozoal agents (Experimental): Combination of two selected anti-protozoal agents with documented anti-cancer properties
  Interventions: Drug: Anti-Protozoal Agents
- Anti-bacterial + anti-fungal + anti-protozoal agents (Experimental): Combination of six selected anti-bacterial agents, anti-fungal agents, and anti-protozoal agents with documented anti-cancer properties
  Interventions: Drug: Anti-Bacterial Agents; Drug: Anti-Fungal Agents; Drug: Anti-Protozoal Agents

INTERVENTIONS:
Drug: Anti-Bacterial Agents — Doxycycline, Paramomycin, Clarithromycin, Clindamycin, Dapsone, Miltefosine
  Arms: Anti-bacterial + anti-fungal + anti-protozoal agents; Anti-bacterial agents
Drug: Anti-Fungal Agents — Itraconazole, Amphotericin B liposomal, Fluconazole, Terbinafine, Voriconazole
  Arms: Anti-bacterial + anti-fungal + anti-protozoal agents; Anti-fungal agents
Drug: Anti-Protozoal Agents — Nitazoxanide, Chloroquine, Albendazole, Ivermectin, Mebendazole, Metronidazole, Praziquantel, Levamisole
  Arms: Anti-bacterial + anti-fungal + anti-protozoal agents; Anti-protozoal agents

SUMMARY:
The cell behavior that the investigators regard as "malignant," including: cell autonomy; invasion and digestion of surrounding normal tissues; migration and colonization of distant organs; ability to develop resistance to drugs, temperature, or radiation; and ability to kill the host, are not only characteristics of cancer cells, but of pathogenic and/or opportunistic unicellular organisms (bacteria, fungi and protozoa). Rudolf Virchow (1821-1902), the father of modern pathology, first pointed out the resemblance between the biological behavior of cancer cells and that of single-celled organisms when causing infections. He thought, incorrectly, that cancer cells were cells infected with bacteria and had acquired their pathogenic behavior from them. Others later postulated that the behavior of cancer cells was likely due to the re-expression of past traits and behaviors (atavism) derived from their past evolutionary experience as independent, single-celled organisms from which all cells in multicellular organisms originated. In other words, the behavior of pathogenic unicellular organisms, including: unlimited replicative potential; capacity for invasion, migration, and metastases; abilities to evade the host's immune system, to generate multi-drug resistance; and to kill a host, are what the investigators define as "cancer" when one of the investigators cells re-express these past ancestral traits. This reversion or de-evolution of a differentiated cell to its ancestral undifferentiated, unicellular form has been named "Atavistic Metamorphosis."

This does not imply that cancer cells are bacteria, protozoa, or yeasts. It means that cancer cells express functions and/or behaviors similar to their ancestral parents, the unicellular organisms from which our cells originated.

If this is true, a combination of drugs that are effective to eradicate certain unicellular organisms may work in cancer treatment.

The principal objective of this study is to determine whether there is a benefit for patients with advanced, metastatic and terminal cancers to be treated with combinations of selected drugs conventionally used in medical practice to kill bacterial, fungal and protozoal cells.

DETAILED DESCRIPTION:
This is an investigator initiated, randomized, single-blind, response-adaptive trial conducted at two sites in patients who have tried conventional therapy and failed or have refused conventional therapy. This study is being conducted to determine the efficacy of combinations of marketed drugs against unicellular organisms in cancer treatment. The products under investigation include FDA- and SSA-approved anti-bacterial, anti-fungal and anti-protozoan drugs with documented anti-cancer properties. The drugs under study are compatible with each other, and used at pharmacological dosages known to be tolerable and safe in humans and/or cancer patients with limited adverse effects. Patients receive treatment for 10 to 12 months. The duration of treatment is depended on the drugs investigated. It is hypothesized that regression will occur within 6 months and treatment will be continued with the assumption that this may prevent recurrences. Outcomes will be measured objectively and assessments appropriate for the type of cancer treated. Outcome measures may include 1) Changes in signs and symptoms; (2) Visual inspection of tumors using weekly photographs and measurements (as appropriate); (3)Monthly chest X-rays to monitor lung tumors, lung metastases and/or fluid in the chest; (4) Ultrasound to evaluate abdominal tumors (e.g., liver metastases), and breast and armpit lymph nodes; (5) CT, MRI and PET scans; (6) Tumor markers in blood such as Carcinoembryonic Antigen (CEA), CA-15.3, CA-19-9, etc. and other laboratory studies to monitor response. The overall goal of this study is to understand the efficacy of atavistic chemotherapy that may mediate metastatic or terminal cancer regression or cure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant disease confirmed histologically that is considered untreatable, progressive and fatal within the next 16 months.
* Patient with an expectation of life greater than 3 months.
* Patients with malignant disease that may be evaluated or measured clinically either through radiographic studies, visually, histologically, in serum or blood tumor markers, or through any other method medical approved for that disease.

Exclusion Criteria:

* Patients over 75 years of age.
* Patients who are pregnant.
* Patients that have a known allergy to any of the drugs planned for use.
* Patients with renal, hepatic, pulmonary, cardiovascular compromise, or other systemic or other clinical conditions such as AIDS, tuberculosis, etc., which, in the opinion of the Investigator, may pose a risk to the subject.
* Malignancies of hemato-lymphatic origin (leukemias and lymphomas)

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2011-07-26 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy as measured by the number of participants with an objective clinical tumor regression response | 6 Months
  Tumor regression will be measrued objectively and assessments appropriate for the type of cancer treated. Outcome measures may include 1) Changes in signs and symptoms; (2) Visual inspection of tumors using weekly photographs and measurements (as appropriate); (3)Monthly chest X-rays to monitor lung tumors, lung metastases and/or fluid in the chest; (4) Ultrasound to evaluate abdominal tumors (e.g., liver metastases), and breast and armpit lymph nodes; (5) CT, MRI and PET scans; (6) Tumor markers in blood such as Carcinoembryonic Antigen (CEA), CA-15.3, CA-19-9 and other laboratory studies to monitor response.

SECONDARY OUTCOMES:
Clinical efficacy as measured by the number of participants with an objective clinical tumor regression response | 12 Months
  Tumor regression will be measrued objectively and assessments appropriate for the type of cancer treated. Outcome measures may include 1) Changes in signs and symptoms; (2) Visual inspection of tumors using weekly photographs and measurements (as appropriate); (3)Monthly chest X-rays to monitor lung tumors, lung metastases and/or fluid in the chest; (4) Ultrasound to evaluate abdominal tumors (e.g., liver metastases), and breast and armpit lymph nodes; (5) CT, MRI and PET scans; (6) Tumor markers in blood such as Carcinoembryonic Antigen (CEA), CA-15.3, CA-19-9 and other laboratory studies to monitor response.
Clinical safety as measured by the incidence of adverse events in each intervention group | 12 Months
  Determine the percentage of incidence of adverse events in each intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Arguello, MD, Principal Investigator — Dr. Frank Arguello Cancer Clinic; Rafael Argüello-Astorga, MD, PhD, Principal Investigator — Instituto de Ciencia y Medicina Genomica
Locations (2):
- Mexico (2):
  - Dr. Frank Arguello Cancer Clinic, San José del Cabo, Baja California Sur
  - Instituto de Ciencia y Medicina Genomica, Torreón, Coahuila

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arguello F, Baggs RB, Frantz CN. A murine model of experimental metastasis to bone and bone marrow. Cancer Res. 1988 Dec 1;48(23):6876-81. PMID 3180096
- [Background] Arguello F, Alexander M, Sterry JA, Tudor G, Smith EM, Kalavar NT, Greene JF Jr, Koss W, Morgan CD, Stinson SF, Siford TJ, Alvord WG, Klabansky RL, Sausville EA. Flavopiridol induces apoptosis of normal lymphoid cells, causes immunosuppression, and has potent antitumor activity In vivo against human leukemia and lymphoma xenografts. Blood. 1998 Apr 1;91(7):2482-90. PMID 9516149
- [Background] Arguello F, Baggs RB, Duerst RE, Johnstone L, McQueen K, Frantz CN. Pathogenesis of vertebral metastasis and epidural spinal cord compression. Cancer. 1990 Jan 1;65(1):98-106. doi: 10.1002/1097-0142(19900101)65:13.0.co;2-k. PMID 2293874
- [Background] Arguello F, Furlanetto RW, Baggs RB, Graves BT, Harwell SE, Cohen HJ, Frantz CN. Incidence and distribution of experimental metastases in mutant mice with defective organ microenvironments (genotypes Sl/Sld and W/Wv). Cancer Res. 1992 Apr 15;52(8):2304-9. PMID 1559233
- [Background] Arguello F, Baggs RB, Graves BT, Harwell SE, Cohen HJ, Frantz CN. Effect of IL-1 on experimental bone/bone-marrow metastases. Int J Cancer. 1992 Nov 11;52(5):802-7. doi: 10.1002/ijc.2910520522. PMID 1428234
- [Background] Arguello F, Sterry JA, Zhao YZ, Alexander MR, Shoemaker RH, Cohen HJ. Two serologic markers to monitor the engraftment, growth, and treatment response of human leukemias in severe combined immunodeficient mice. Blood. 1996 May 15;87(10):4325-32. PMID 8639792
- See also: STAGE IV MELANOMA PATIENTS TREATED WITH ATAVISTIC CHEMOTHERAPY — http://atavisticchemotherapy.com/wp-content/uploads/2017/11/ENGLISHMELANOMA_CASES.pdf
- See also: STAGE IV BREAST CANCER PATIENTS TREATED WITH ATAVISTIC CHEMOTHERAPY — http://atavisticchemotherapy.com/wp-content/uploads/2017/11/ENGLISHBREASTCANCER_CASES.pdf
- See also: What is Atavistic Chemotherapy? — https://www.youtube.com/watch?v=KwX43KPbpDY
- See also: Website Atavistic Chemotherapy — http://www.atavisticchemotherapy.com
- See also: Facts of Evolution — https://www.youtube.com/watch?v=nvJFI3ChOUU